CLINICAL TRIAL: NCT01192373
Title: Short Term Modulation of Circulating Free Fatty Acids in Heart Failure Patients With Type 2 Diabetes: "Effect on Myocardial Lipid Content, Left Ventricular Function and Exercise Capacity"
Brief Title: Modulation of Free Fatty Acids in Heart Failure Patients With Diabetes: "Effect on Left Ventricular Function"
Acronym: Metamod3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M20090230
Record Dates: First submitted 2010-08-24; First posted 2010-09-01 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Heart Failure; Diabetes
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High circulating free fatty acids (Experimental): using Heparin af intralipid infusion for 8 hours
  Interventions: Other: Metabolic substrate modulation
- Low circulation free fatty acids (Active Comparator): using hyperinsulinaemic euglycemic clamp for 8 hours
  Interventions: Other: metabolic substrate modulation

INTERVENTIONS:
Other: Metabolic substrate modulation — for high circulation free fatty acids: Heparin (250IE/hour) + intralipid (20%, 62 ml/hour).
  Arms: High circulating free fatty acids
Other: metabolic substrate modulation — low circulating free acids: hyperinsulinaemic euglycemic clamp (0,8 mUkg/min) with venous blood glucose at 4,5-6,5 mM.
  Arms: Low circulation free fatty acids

SUMMARY:
The investigators wish to investigate the the short term effect of low circulating free fatty acids in congestive heart failure patients with type 2 diabetes.

Hypothesis: Low levels of circulating free fatty acids decrease myocardial and peripheral muscle lipid content, improves cardiac performance and exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* ejection fraction at or lower than 45%
* type 2 diabetes

Exclusion Criteria:

* known s-creatinine >220mM
* known S-alanine aminotransferase >3 times normal upper limit
* other disabilitating conditions
* pregnancy
* insulin treatment

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Left ventricular function | 1-6 weeks
  Left ventricular systolic function (Ejection fraction, tissue velocity, Strain and strain rate).
  Left ventricular diastolic funtion (E/A ratio, E/e' ratio, IVRT) Cardiac output. All parameters measured at rest and peak exercise and outcome is difference between low and high ciculating free fatty acids.
intracellular lipid content | 1-6 weeks
  Magnetic Resonans proton spectroscopy (septal myocardial intracellular lipid content) Magnetic Resonans proton spectroscopy (Tibialis anterior muscle intracellular lipid content).
  Outcome is difference between low and high ciculating free fatty acids.
Exercise capacity and oxygen consumption | 1-6 weeks
  Using treadmill and continues oxygen consumption measurement. Outcome is difference between low and high ciculating free fatty acids.

SECONDARY OUTCOMES:
Regional left ventricular function | 1-6 weeks
  regional speckle tracking during rest and peak exercise. Outcome is difference between low and high ciculating free fatty acids.
6 minutes hall walk test | 1-6 weeks
  distance difference between low and high levels of circulating FFA. Outcome is difference between low and high ciculating free fatty acids.
metabolic and hormonal profile | 1-6 weeks
  bloodsamples

CONTACTS AND LOCATIONS:
Overall Officials: Roni R Nielsen, MD, Principal Investigator — Dept. of cardiolgy, Aarhus University hospital, Skejby. Brendstrupgaardsvej 100, 8200 Aarhus N, Denmark
Locations (1):
- Dept. of cardiology, Aarhus University hospital Skejby,, Aarhus, Region Midjylland, Denmark

REFERENCES:
- [Derived] Nielsen R, Norrelund H, Kampmann U, Kim WY, Ringgaard S, Schar M, Moller N, Botker HE, Wiggers H. Failing heart of patients with type 2 diabetes mellitus can adapt to extreme short-term increases in circulating lipids and does not display features of acute myocardial lipotoxicity. Circ Heart Fail. 2013 Jul;6(4):845-52. doi: 10.1161/CIRCHEARTFAILURE.113.000187. Epub 2013 Jun 3. PMID 23733915